CLINICAL TRIAL: NCT05313750
Title: Efficacy and Safety of Sitafloxacin in the Treatment of Acute Exacerbation of Bronchiectasis in Adults :A Multi-center, Randomized, Evaluator-blinded, Levofloxacin Parallel-controlled Clinical Study
Brief Title: Efficacy and Safety of Sitafloxacin in the Treatment of Acute Exacerbation of Bronchiectasis in Adults
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Jin-Fu Xu, Chief of Department of Pulmonary and Critical Care Medicine, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20211112
Record Dates: First submitted 2021-11-12; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Acute Exacerbation of Bronchiectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sitafloxacin group (Experimental): Oral sitafloxacin (0.1g one time daily) for 10 days
  Interventions: Drug: anti-infective therapy sitafloxacin
- levofloxacin group (Active Comparator): Oral levofloxacin (0.4g one time daily) for 10 days
  Interventions: Drug: anti-infective therapy levofloxacin

INTERVENTIONS:
Drug: anti-infective therapy sitafloxacin — anti-infective therapy
  Arms: sitafloxacin group
Drug: anti-infective therapy levofloxacin — anti-infective therapy
  Arms: levofloxacin group

SUMMARY:
The treatment of acute exacerbation of bronchiectasis requires comprehensive treatment, and antibacterial drug therapy is the key. The study is a multicenter, randomized, evaluator-blinded, levofloxacin parallel-controlled clinical study designed to evaluate the efficacy and safety of sitafloxacin in the treatment of acute exacerbations of bronchiectasis in adults.

DETAILED DESCRIPTION:
Acute exacerbation of bronchiectasis refers to changes in three or more ofthe following six symptoms in patients with bronchiectasis, including cough frequency, increased sputum volume or nature change, increased purulent sputum with or without wheezing, dyspnea, hemoptysis, and (or) general malaise, lasting for 48 hours or more, and clinicians consider that it is necessary to change the current therapeutic regimen for the condition. The treatment of acute exacerbation of bronchiectasis requires comprehensive treatment, and antibacterial drug therapy is the key. Sitafloxacin has a broad antibacterial spectrum. It has good in vivo and in vitro activities against gram-positive bacteria, gram-negative bacteria, anaerobic bacteria and atypical pathogens and it has excellent pharmacokinetic properties, rapid oral absorption, strong tissue permeability and no liver retention, and no inhibition to main liver drug enzymes of human and it shows good activity against many fluoroquinolone-resistant bacteria. The study aims to evaluate efficacy and safety of sitafloxacin in the treatment of acute exacerbations of bronchiectasis in adults.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who older than 18 years old and are diagnosed with acute exacerbations of bronchiectasis Acute exacerbation of bronchiectasis refers to changes in three or more ofthe following six symptoms in patients, including cough frequency, increased sputum volume or nature change, increased purulent sputum with or without wheezing, dyspnea, hemoptysis, and (or) general malaise, lasting for 48 hours or more, and clinicians consider that it is necessary to change the current therapeutic regimen for the condition; It should also be noted that left and right cardiac insufficiency, arrhythmia, pleural effusion, pulmonary embolism, pneumothorax and pneumonia should be noted.
2. Patients who have not accepted antibacterial drug therapy within 48 hours before initiation of administration or who have accepted other antibacterial drug therapy within 48 hours before initiation of administration but not more than 24 hours (excluding use of quinolones), and still present with apparent symptoms of infection

Exclusion Criteria:

Patients complying with any of the following exclusion criteria cannot be enrolled into this trail:

1. Bronchiectaticpatientswith previous sputum examinations suggesting the presence of bronchiectasis of pathogenic

   - Page 3 of 5 - microorganisms resistant to quinolone drugscomplicated with chronic respiratory failure
2. Patients with a previous stable phase BSI score greater than 9
3. Inhaled, oral or intravenous quinolone antibiotics have been used within 1 week before enrollment.
4. Patients who have a history of allergy to any quinolone or fluoroquinolone
5. Patients who have a medical history of pathological changes in the muscle tendon caused by quinolones or fluoroquinolones;
6. Complicatingbronchial asthma, allergic bronchopulmonary aspergillosis, or active tuberculosis, or active non-tuberculous mycobacterial infection that requires standardized treatment;
7. A history of complicating serious cardiovascular diseases, hematopoietic system diseases, etc. (such as: congestive heart failure, clinically significant coronary heart disease, stroke, myocardial infarction and/or stroke that occurred within half a year, clinically significant arrhythmia, known aortic aneurysm, poorly controlled hypertension (systolic blood pressure> 160mmHg, or diastolic blood pressure> 100mmHg, etc.in two or more consecutive detections);
8. Moderate hemoptysis (>30ml in 24h);
9. Complicatingserious systemic diseases and mental disorders;
10. Complicatingdiabetic patients with poor control or fasting blood glucose> 10mmol/L;
11. Complicatingmalignant tumor;
12. Complicating myasthenia gravis and Parkinson's disease;
13. Patients with abnormal liver function test, withAST (GOT) and/or ALT (GPT) higher than 3 times the upper limit of normal, and/or total bilirubin higher than twice the upper limit of normal;
14. Patients with moderate or severe renal hypofunction, withendogenous creatinine clearance rate <50 ml/min (if the examination is not performed, the clearance rate may be calculated from the serum creatinine value using a formula)*;
15. *Cockcroft-Gault Formula i. Male:eCcr(ml/min)=[(140 - age)

    ×weight(kg)]/[72 ×serum creatinine(mg/dl)] ii. Female:eCcr(ml/ min)=[(140 - age) ×weight(kg) × 0.85]/[72 ×serum creatinine(mg/ dl)] or, iii. Male: eCcr(ml/min)= [(140 - age)×weight(kg)×1.23]/serum creatinine(µmol/l) iv. Male:eCcr(ml/min)= [(140 - age)×weight× 1.04]/serum creatinine(µmol/l)
16. Patients with a medical history of prolonged QTc interval,or requiring use of drugs to treat prolonged QTc interval (e.g., Class I or III anti-arrhythmic, as detailed in Appendix 1), or suffering serious cardiac insufficiency (NYHA Functional Class ≥ III, as detailed in Appendix 2);
17. Patients with a medical history of epileptic seizures, or mental disease that may influence the compliance withthe protocol, or with suicide risk, or a history of alcohol or illicit drug abuse;
18. Immunocompromised patients usingglucocorticoids (with the total dose equivalent to prednisone daily or acourse of treatment of more than 2 weeks) or immunosuppressants, etc.;
19. Pregnant or lactating women or women of childbearing age who are preparing to conceive;
20. Those who have participatedin other clinical trials within 3 months prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical effectiveness | 24days
  The clinical effective rate was the percentage of improved cases in the analysis set cases.

SECONDARY OUTCOMES:
microbiological discontinuation of Administration | 10days
  The effective rate of microbiology is the percentage of cases of clearance, hypothetical clearance, replacement and reinfection in the number of evaluable cases in the analysis set.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai pulmonary hospital, Shanghai, Shanghai Municipality, China